CLINICAL TRIAL: NCT05525676
Title: Supporting Relationships to Reduce Suicide Risk: A Randomized Control Trial of the Brief Relationship Checkup
Brief Title: Relationship Checkups to Reduce Veteran Suicide Risk
Acronym: BRC RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3823-W; IK2RX003823 (NIH)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Relationship Distress; Mental Health
Keywords: Randomized Controlled Trial; Couple therapy; Primary Care; Partner Communication
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial design. Participants in both arms will receive active treatments that are matched for length (three, 30-minute sessions) over a 45 day period. After that couples will be assessed for 6 months.
Who Masked: Outcomes Assessor
Masking Description: The interviewer who evaluates clinical outcomes will not know the assigned condition of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief Relationship Checkup (BRC) (Experimental): Couples in the experimental condition will participate in three joint sessions of the Brief Relationship Checkup (BRC; Cordova 2014; Cigrang et al., 2016). This program has been tested in Air Force Primary Care but has not been explored in Veterans with ongoing mental health issues and has not been compared to an active treatment.
  Interventions: Behavioral: Brief Relationship Checkup (BRC)
- Co-Located Collaborative Care (CCC) (Active Comparator): The comparison condition will be three sessions of Co-Located Collaborative Care (CCC) offered to the Screened Veteran only. This reflects the current standard of care in VA Primary Care Mental Health.
  Interventions: Behavioral: Co-Located Collaborative Care (CCC)

INTERVENTIONS:
Behavioral: Brief Relationship Checkup (BRC) — The investigators are using the three 30-minute session protocol developed for Air Force Primary Care (Cigrang et al., 2016). Although it is simply referred to as the "Marriage Checkup" in that manuscript, the investigators use the name BRC to distinguish it from many other versions of Dr. James Cordova's Marriage Checkup (Cordova, 2014) adapted for different settings. Sessions in this version are briefer than other versions (30 mins vs. 60-90 mins) and this trial does not have any eligibility restrictions based on marital status.
  Other Names: Marriage Checkup; Relationship Checkup
  Arms: Brief Relationship Checkup (BRC)
Behavioral: Co-Located Collaborative Care (CCC) — The investigators are using the Co-Located Collaborative Care model developed by the VA Center for Integrated Healthcare to deliver at all VAs. Although the CCC model is flexible and can range from 1-6 sessions, in this study the investigators standardize the model to three sessions for a clear comparison with BRC. Session 1 uses the CCC "Functional Assessment"/"Initial Assessment" protocol. Sessions 2 & 3 use the CCC Follow-up protocol.
  Session 1 (25-30 min)- Veteran completes a functional assessment of concerns (15 mins) and then develops a personalized action plan (10 minutes) Session 2 (25-30 min)- Veteran's progress addressing concerns is assessed (5 mins) and the remainder of the session is spend updating the action plan (20 minutes) Session 3 (25-30 min)- Veteran's progress addressing concerns is assessed (5 mins) and the remainder of the session is spend updating the action plan, including receiving referrals (20 minutes)
  Other Names: Behavioral Health Consultation
  Arms: Co-Located Collaborative Care (CCC)

SUMMARY:
This study compares two approaches to working with Veterans that have a mix of mental health and relationship concerns in primary care. One approach is a 3-session couple-based program called the Brief Relationship Checkup (BRC). BRC has shown promise improving relationship health in Air Force primary care (including some mental health symptoms related to relationship functioning) but has never been tested for individuals with significant mental health concerns. The other approach is a high-quality delivery of three sessions of Co-Located Collaborative Care (CCC) with the Screened Veteran only. This program is the current standard of care for Veterans reporting mental health concerns in primary care (including mental health concerns related to their relationship) but has never been tested for individuals struggling with relationship concerns. The goal is to compare the benefits of the couples-based program vs. the individual-based program when it comes to reducing suicide risk factors at the relationship level and the individual level.

DETAILED DESCRIPTION:
BACKGROUND: Romantic relationship distress is a common area of concern for Veterans struggling with depression, posttraumatic stress disorder (PTSD), alcohol misuse, and suicide ideation. In a study of Veterans who screened positive for the above concerns in primary care, 58% of partnered Veterans reported romantic relationship problems. Relationship problems are also a prominent risk factor for suicide, preceding 24% of Veteran suicide deaths and 50% for Veterans 18-35. Conversely, full participation in mutually supportive relationships confers protection against suicide. This suggests it may be able to offset risk by turning distressed relationships into protective partnerships. Unfortunately, the intensive formats of existing couple therapies result in couples discontinuing after 2-3 sessions or delaying treatment until they are close to breakup. This underscores the need for brief relationship support that is accessible through primary care mental health (PC-MHI).

Relationship Checkup programs incorporates a combination of couple therapy and motivational interviewing techniques to encourage couples to make concrete commitments to improve their relationship. The Brief Relationship Checkup (BRC) is a three 30-minute session version initially designed to address relationship distress in primary care. BRC demonstrates efficacy in reducing suicide risk factors such as relationship dysfunction and depressed mood while promoting protective factors such as mutual responsiveness to one another's concerns, a core element of supportive relationships. Earlier Checkup programs have also been shown to increase individual and couple therapy engagement. In an open label pilot trial, the investigators found BRC was feasible and acceptable to Veterans screening positive on VA PC-MHI screens. The investigators also found its highly structured framework could be learned by trainees without prior couple therapy experience.

RESEARCH PLAN: This study is a randomized controlled trial (RCT) of BRC administered to evaluate its ability to modify suicide risk/protective factors. Up to 360 participants will be enrolled and screened by phone to identify couples that are in distressed committed relationship where at least one partner is a Veteran who screens positive on a PC-MHI screen for common suicide risk factors including suicide ideation, depression, PTSD, or alcohol misuse (the "Screened Veteran"). The target is to randomize 72 couples (144 individuals) to BRC or to three sessions of the current PC-MHI Co-Located Collaborative Care model (CCC) for the Screened Veteran only. All participants will complete baseline, post-treatment, 3-month, and 6-month assessments.

SPECIFIC AIMS: The study will provide the foundations for a larger clinical trial proposal through pursuit of the following research aims and hypotheses (H):

AIM 1: Determine BRC's efficacy in improving relationship factors related to suicide for both partners.

AIM 2: Determine BRC's efficacy in improving individual factors related to suicide for the Screened Veteran.

AIM 3: Develop and validate a fidelity codebook to operationalize BRC adherence and clinician competency.

ELIGIBILITY:
Inclusion Criteria:

1. BOTH PARTNERS must be age 18 or over
2. BOTH PARTNERS must demonstrate sufficient knowledge of English and cognitive capacity to understand the study through comprehension of consent questions
3. BOTH PARTNERS must self-identify as "in a committed relationship" with their partner for at least 6-months.
4. AT LEAST ONE PARTNER must report at least mild relationship distress on a relationship satisfaction screen (CSI-4).
5. AT LEAST ONE PARTNER must be a VHA-enrolled Veteran who screens positive on a VA Primary Care Mental Health Screen for ONE OR MORE of the following conditions: Depressed Mood, Unsafe drinking, Posttraumatic stress, or Suicidal Ideation.

Exclusion Criteria:

1. EITHER PARTNER reports that they are already engaged in ongoing couple or family therapy.
2. EITHER PARTNER reports severe intimate partner violence in the last year.
3. EITHER PARTNER reports ongoing or upcoming legal conflicts between one another (e.g., custody dispute; restraining order; divorce proceedings)
4. EITHER PARTNER reports experiencing suicidal intent requiring hospitalization.
5. EITHER PARTNER experiences past-month psychosis or mania.
6. EITHER PARTNER has completed therapy with the PI, Dr. Dev Crasta, within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Relationship Functioning | Change from Baseline (First Assessment) to Post-Treatment (approx. 1.5 months after randomization)
  Relationship Functioning will be measured using the Couples Satisfaction Index (CSI). The self-report scale has a minimum of 0 and a maximum of 161 with higher scores representing more satisfying relationships and scores < 104.5 classified as "distressed." The CSI is widely used in couple therapy research and is used routinely in VA care to evaluate Veterans' progress in evidence-based couple therapies. Analyses will compare relationship functioning across both Screened Veterans and their Partners using 3-level multilevel models with waves of assessment (Level 1) nested within individual partners (Level 2) nested within couples (Level 3). Treatment efficacy is defined as the gains in satisfaction being significantly greater in one arm than the other (p<.05).
Relationship Functioning | Monthly Change over 6 Months Post-Treatment (approx. 1.5 months to 7.5 months after randomization)
  Relationship Functioning will be measured using the Couples Satisfaction Index (CSI). The self-report scale has a minimum of 0 and a maximum of 161 with higher scores representing more satisfying relationships and scores < 104.5 classified as "distressed." The CSI is widely used in couple therapy research and is used routinely in VA care to evaluate Veterans' progress in evidence-based couple therapies. Analyses will compare relationship functioning across both Screened Veterans and their Partners using 3-level multilevel models with waves of assessment (Level 1) nested within individual partners (Level 2) nested within couples (Level 3).

SECONDARY OUTCOMES:
Emotional Intimacy/Mutual Responsiveness | Change from Baseline (First Assessment) to Post-Treatment (approx. 1.5 months after randomization)
  Emotional Intimacy will be measured using the Perceived Responsiveness & Insensitivity Scale (PRI). The PRI has a minimum of 0 and a maximum of 80. The PRI is an optimized measure of "Perceived Partner Responsiveness," a model of emotional intimacy that is widely used in the field to understand whether partners see one another as understanding/caring. Analyses will compare responsiveness across both Screened Veterans and their Partners using 3-level multilevel models with waves of assessment (Level 1) nested within individual partners (Level 2) nested within couples (Level 3). Treatment efficacy is defined as the gains in intimacy being significantly greater in one arm than the other (p<.05).
Emotional Intimacy/Mutual Responsiveness | Monthly Change over 6 Months Post-Treatment (approx. 1.5 months to 7.5 months after randomization)
  Emotional Intimacy will be measured using the Perceived Responsiveness & Insensitivity Scale (PRI). The PRI has a minimum of 0 and a maximum of 80. The PRI is an optimized measure of "Perceived Partner Responsiveness," a model of emotional intimacy that is widely used in the field to understand whether partners see one another as understanding/caring. Analyses will compare responsiveness across both Screened Veterans and their Partners using 3-level multilevel models with waves of assessment (Level 1) nested within individual partners (Level 2) nested within couples (Level 3).
Treatment Engagement in Mental Health Services | 180 day period after Post-Treatment session (1.5 months after randomization)
  Treatment engagement in mental health services will be assessed through a review of the electronic medical record over each of the following windows: 1) 180-day period prior to baseline session; 2) during the treatment period from baseline to post-treatment, 3) the 180-day period after the post-treatment assessment. Over each window, staff will review appointments (e.g., individual, group, assessments), consults placed (e.g., General Mental Health; MST coordinator); and new prescriptions. Analyses will compare treatment engagement using 2-level multilevel models with assessment periods (Level 1) nested within Screened Veterans (Level 2). Their partners may or may not have VA electronic medical records, but available partner data will be used as a covariate. Treatment efficacy is defined as the Screened Veterans' treatment engagement being significantly greater in one arm than the other after accounting for treatment utilization prior to baseline (p<.05).

OTHER OUTCOMES:
Depressive Symptoms | Change from Baseline (First Assessment) to Post-Treatment (approx. 1.5 months after randomization)
  Depression will be measured using the 9-item Patient Health Questionnaire (PHQ-9). This self-report scale has a minimum of 0 and a maximum of 27 with higher scores representing greater number and frequency of depression symptoms and scores of 10 or higher representing moderate depression. Exploratory analyses will calculate 95% confidence intervals to compare Screened Veteran trajectories across the two study arms.
Posttraumatic Stress Disorder (PTSD) Symptom Severity | Change from Baseline (First Assessment) to Post-Treatment (approx. 1.5 months after randomization)
  Posttraumatic symptom will be measured using the Posttraumatic Stress Disorder Checklist for the DSM-5 (PCL-5). This self-report scale has a minimum of 0 and a maximum of 80 with higher scores representing more extreme symptoms and scores of 33 or higher representing probable PTSD. The PCL-5 is used routinely in VA care to evaluate Veterans' progress in long-term PTSD treatment. Exploratory analyses will calculate 95% confidence intervals to compare Screened Veteran trajectories across the two study arms.
Depressive Symptoms | Monthly Change over 6 Months Post-Treatment (approx. 1.5 months to 7.5 months after randomization)
  Depression will be measured using the 9-item Patient Health Questionnaire (PHQ-9). This self-report scale has a minimum of 0 and a maximum of 27 with higher scores representing greater number and frequency of depression symptoms and scores of 10 or higher representing moderate depression. Exploratory analyses will calculate 95% confidence intervals to compare Screened Veteran trajectories across the two study arms.
Posttraumatic Stress Disorder (PTSD) Symptom Severity | Monthly Change over 6 Months Post-Treatment (approx. 1.5 months to 7.5 months after randomization)
  Posttraumatic symptom will be measured using the Posttraumatic Stress Disorder Checklist for the DSM-5 (PCL-5). This self-report scale has a minimum of 0 and a maximum of 80 with higher scores representing more extreme symptoms and scores of 33 or higher representing probable PTSD. The PCL-5 is used routinely in VA care to evaluate Veterans' progress in long-term PTSD treatment. Exploratory analyses will calculate 95% confidence intervals to compare Screened Veteran trajectories across the two study arms.
Alcohol Use | Change from Baseline (First Assessment) to Post-Treatment (approx. 1.5 months after randomization)
  Alcohol use over the study will be monitored using a 30-day "Timeline Follow Back" protocol (TLFB). In this "semi-structured interview," the interviewer helps participants recollect on which days they drank and how many drinks they had each day. Exploratory analyses will calculate 95% confidence intervals to compare Screened Veteran trajectories across the two study arms.
Alcohol Use | Monthly Change over 6 Months Post-Treatment (approx. 1.5 months to 7.5 months after randomization)
  Alcohol use over the study will be monitored using a 30-day "Timeline Follow Back" protocol (TLFB). In this "semi-structured interview," the interviewer helps participants recollect on which days they drank and how many drinks they had each day. Exploratory analyses will calculate 95% confidence intervals to compare Screened Veteran trajectories across the two study arms.
Suicide Ideation Severity | Change from Baseline (First Assessment) to Post-Treatment (approx. 1.5 months after randomization)
  Suicide ideation over the study will be monitored using the "Last Month" version of the Columbia Suicide Severity Rating Scale (CSSRS). This semi-structured interview has interviewers rate suicide ideation on a scale of 0 to 5, with scores of 3-5 placing individuals at high risk for attempt. VA hospitals use the C-SSRS across all clinics. In cases where participants miss an assessment, the investigators will review the chart to identify a C-SSRS close to the target date. Exploratory analyses will calculate 95% confidence intervals to compare Screened Veteran trajectories across the two study arms.
Suicide Ideation Severity | Monthly Change over 6 Months Post-Treatment (approx. 1.5 months to 7.5 months after randomization)
  Suicide ideation over the study will be monitored using the "Last Month" version of the Columbia Suicide Severity Rating Scale (CSSRS). This semi-structured interview has interviewers rate suicide ideation on a scale of 0 to 5, with scores of 3-5 placing individuals at high risk for attempt. VA hospitals use the C-SSRS across all clinics. In cases where participants miss an assessment, the investigators will review the chart to identify a C-SSRS close to the target date. Exploratory analyses will calculate 95% confidence intervals to compare Screened Veteran trajectories across the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Dev J Crasta, Principal Investigator — VA Finger Lakes Healthcare System, Canandaigua, NY
Locations (1):
- VA Finger Lakes Healthcare System, Canandaigua, NY, Canandaigua, New York, United States

IPD SHARING:
Plan to Share IPD: No